CLINICAL TRIAL: NCT03804424
Title: Early Phase I Evaluation of 64Cu-LLP2A for Imaging Multiple Myeloma
Brief Title: 64Cu-LLP2A for Imaging Multiple Myeloma
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Drug formulation changed, opening new trial
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Diagnostic
Other Study IDs: 201807197
Record Dates: First submitted 2018-12-10; First posted 2019-01-15 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Blood Specimen Collection; Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Images will be assessed by independent observers (nuclear medicine expert in evaluating PET images using novel radiotracers, and MR radiologist expert in evaluating MR images), who will initially be blinded to all clinical information available (such as tumor size and location), which will be followed by un-blinded combined reading of the PET and MR images
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1: Pilot 64Cu-LLP2A Imaging (Experimental): * 16 adult individuals (6-8 patients with known MM; 6-10 healthy volunteers)
  * All subjects who enter the study in Cohort 1 will be injected with up to 11 mCi of 64Cu-LLP2A and will undergo body imaging at least twice within 0-30 hrs following administration of 64Cu-LLP2A to study tracer biodistribution and calculate human dosimetry
  * 6 subjects will also undergo dynamic study for 60 mins immediately after administration of 64Cu-LLP2A.
  Interventions: Drug: 64Cu-LLP2A; Device: PET/MR; Procedure: Blood samples for serum stability; Procedure: Blood samples for metabolite analysis; Procedure: Urine sample; Procedure: Electrocardiogram; Device: PET/CT
- Cohort 2: Quantitative 64Cu-LLP2A Imaging (Experimental): * 20 patients with MM will be recruited
  * Subjects who enter on study in Cohort 2 will undergo a 60-min dynamic imaging over the known site of disease (OR pelvis and lower lumbar spine, if no site of disease is known). Following a simple DIXON MRI or low dose CT scan for attenuation correction, subjects will be injected with a dose of up to11 mCi of 64Cu-LLP2A and a list mode dynamic imaging acquisition will begin for a total of 60 mins. Following the dynamic study, or at the optimal time point determined from cohort 1 imaging, after a simple DIXON or low dose CT scan for body (top of the head to below the knees) attenuation correction, emission scans (2-5 min per bed position) will be performed
  Interventions: Drug: 64Cu-LLP2A; Device: PET/MR; Procedure: Blood samples for serum stability; Procedure: Blood samples for metabolite analysis; Procedure: Tumor biopsy; Procedure: Electrocardiogram; Device: PET/CT

INTERVENTIONS:
Drug: 64Cu-LLP2A — -64Cu-LLP2A, will be manufactured following batch production record at the cyclotron GMP facility (Washington University School of Medicine GMP radiochemistry/cyclotron facility)
Device: PET/MR — -All PET imaging will be performed as PET/MR or PET/CT
Procedure: Blood samples for serum stability — -3 venous samples obtained from an IV site separate from the site of 64Cu-LLP2A injection (2 mL each) will be obtained at the following time points: Cohort 1: prior to injection, at completion of dynamic scanning in those who undergo dynamic imaging and at completion of one of the body imaging time points. In those who do not undergo dynamic imaging, prior to injection, and after completing body imaging at 2 of the 3 time points. Cohort 2: subjects will have samples drawn prior to injection, at completion of dynamic scanning, and at completion of body imaging.
Procedure: Blood samples for metabolite analysis — -Typically, 2 blood samples obtained from an IV site separate from the site of 64Cu-LLP2A injection (preferably 1 within the first 5 min and 1 at the completion of the first hour of imaging) will be obtained.
Procedure: Urine sample — -Cohort 1 only
  Arms: Cohort 1: Pilot 64Cu-LLP2A Imaging
Procedure: Tumor biopsy — -Cohort 2 only and only if there hasn't been a recent biopsy of disease
  Arms: Cohort 2: Quantitative 64Cu-LLP2A Imaging
Procedure: Electrocardiogram — -A standard 12-lead ECG will be obtained on all subjects at baseline (within 30 mins prior to injection of 64Cu-LLP2A), and at least 60 minutes post injection or prior to study discharge
  Other Names: ECG
Device: PET/CT — -All PET imaging will be performed as PET/MR or PET/CT

SUMMARY:
The investigators are performing a trial with goals to demonstrate the feasibility of imaging multiple myeloma (MM) patients with 64Cu-LLP2A-positron emission tomography (PET)/magnetic resonance (MR). The investigators suggest that 64Cu-LLP2A will allow for an accurate molecular imaging of MM lesions, which will have an important impact on early stage disease detection and in the long term on the initiation and choice of therapy in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 18 years of age or older with clinically or pathologically defined MM in accordance with International Myeloma Working Group or as stated in office note / clinical assessment from treating physician.

  *All types of active myeloma are eligible including both newly diagnosed and previously treated provided plans are to start a new treatment or restart a prior treatment.
* Healthy Volunteer Subjects: Adult 18 years of age or older with no known hematologic disorder such as anemia, leukemia, etc. who is considered healthy based on assessment by PI. (Cohort 1 only).
* Able to give informed consent.
* Does not have any exclusions related to PET/MR imaging: No implanted medical devices such as: pacemaker, defibrillator, neurostimulator, artificial heart valve, cerebral aneurysm clips, no accidental exposure to metal fragments (if applicable)
* If applicable for administration of contrast with MRI imaging subject must have a calculated GFR of at least 60 mg/mL/1.73 m^2.
* Not currently pregnant or nursing: Subject must be surgically sterile (has had a documented bilateral oophorectomy and/or documented hysterectomy), post-menopausal (cessation of menses for more than 1 year), non-lactating, or of childbearing potential for whom a urine pregnancy test (with the test performed within the 24 hour period immediately prior to administration of 64Cu-LLP2A) is negative.

Exclusion Criteria:

* Patients with other invasive malignancies, with the exception of non-melanoma skin cancer, who had (or have) any evidence of the other cancer present within the last 5 years.
* Unable to tolerate up to 90 min of PET/MR or PET/CT imaging per imaging session.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of imaging MM patients with 64Cu-LLP2A-PET/MR as measured by average organ activity concentration of 64Cu-LLP2A | Up to 30 hours after imaging
  -Average organ activity concentration will be measured and decay corrected by utilizing regions of interest (ROIs) drawn around all organs visible on 64Cu-LLP2A images. Activity organ residence times will be calculated by numerical or analytical integration of the time-activity curves. Uptake/clearance functional fits of mono or bi-exponential functions will be performed and analytical integration, accounted for physical delay, will be performed. The calculated residence times will be used with the program OLINDA/EXM for 64Cu and using the adult human (male/femal) model to calculate the individual organ radiation dose, the whole-body dose, and the effective dose
Feasibility of imaging MM patients with 64Cu-LLP2A-PET/MR as measured by the number of participants who experience an adverse event related to 64Cu-LLP2A | Through 48 hours after last administration of 64Cu-LLP2A (estimated to be at most 4 days)
  -The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for all toxicity reporting.
Feasibility of imaging MM patients with 64Cu-LLP2A-PET/MR as measured by the optimal image time after injection of 64Cu-LLP2A | Up to 30 hours after imaging
  -The optimal imaging time after injection yields the best image quality and tumor-to-non-tumor ratio for visual and quantitative analysis of the lesions
Feasibility of imaging MM patients with 64Cu-LLP2A-PET/MR as measured by image quality of 64Cu-LLP2A-PET/MR images | Up to 30 hours after imaging
  * Overall PET image quality will be graded visually (using 4-point scale with 1 being the worst and poor quality, not acceptable for diagnostic interpretation and 4 being good image quality, similar to routine clinical studies).
  * The images will be assessed by independent observers (a nuclear medicine expert in evaluating PET images using novel radiotracers, and a MR radiologist expert in evaluating MR images
  * The images will then be correlated to MRI (and biopsy if available) to assess whether the lesions identified on 64Cu-LLP2A correspond to myeloma lesions
Feasibility of imaging MM patients with 64Cu-LLP2A-PET/MR as measured by lesion detection of 64Cu-LLP2A-PET/MR images | Up to 30 hours after imaging
  -Lesion detection is measured by lesion uptake in comparison with the surrounding tissue

SECONDARY OUTCOMES:
Comparison of tumor burden (SUVmax) of 64Cu-LLP2A to clinical stage | Up to 30 hours after imaging
  -SUVmax is a mathematical measurement of tumor burden seen on images and calculated by the following equation SUVmax= r / (a'/w) where r= radioactivity concentration in tumor (kBq/ml) as measured by the PET scanner within a defined region of interest, a'=the decay corrected amount of injected 64Cu-LLP2A and w= weight of the patient in grams When PET imaging shows uptake of 64Cyu-LLP2A in site(s) of known tumor the SUVmax will be compared to overall clinical stage as a way to compare accuracy of imaging to known clinical stage
Comparison of tumor burden (SUVmax) of 64Cu-LLP2A to clinical tumor measurement of tumor burden as measured by M-protein of myeloma | Up to 30 hours after imaging
  SUVmax is a mathematical measurement of tumor burden seen on images and calculated by the following equation SUVmax= r / (a'/w) where r= radioactivity concentration in tumor (kBq/ml) as measured by the PET scanner within a defined region of interest, a'=the decay corrected amount of injected 64Cu-LLP2A and w= weight of the patient in grams When PET imaging shows uptake of 64Cyu-LLP2A in site(s) of known tumor the SUVmax will be compared to clinical measurement of tumor burden as seen by the laboratory values for M-protein (lab measurement for myeloma gamma globulin which is increased in multiple myleom due to an abnormal monoclonal proliferation of plasma cells)
Comparision of tumor burden (SUVmax) of 64Cu-LLP2A to clinical measurement of tumor burden as measured by the plasma cell fraction within the bone marrow | Up to 30 hours after imaging
  * Hierarchical models will be used to estimate the correlation of SUVmax with M-protein expression
  * Variance components models will be fit to identify component (proportion) of total variance

CONTACTS AND LOCATIONS:
Overall Officials: Farrokh Dehdashti, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
* A primary means of sharing data will be through publication in peer-reviewed journals. As required by the NIH Public Access Policy, the investigators will submit to the NIH National Library of Medicine's PubMed Central an electronic version of final manuscripts upon acceptance for publication, resulting from research supported by these funds, in whole or in part, with direct costs from NIH.
  * It is expected that approximately 1-2 presentations at national meetings
  * Early phase I evaluation of 64Cu-LLP2A for imaging multiple myeloma will generate imaging, safety and dosimetry data from PET/CT and MR studies of 64Cu-LLP2A. Serum markers such as M-protein, plasma cell density and immunohistochemistry will be correlated with imaging, in order to understand the interaction of 64Cu-LLP2A with VLA-4 in vivo. It is the explicit intention that these data will be placed in a readily accessible public database.
Supporting Information: Study Protocol
Time Frame: All efforts will be made to rapidly release data through publications of the results as quickly as it is possible to analyze the experiments.

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu